CLINICAL TRIAL: NCT03118570
Title: A Phase 2b, Multicentre, Multinational, Double-blind, Dose-finding Study, Incorporating an Open Label Substudy, in Adult Patients With Type I, III or IV Osteogenesis Imperfecta Treated With Setrusumab (BPS804)
Brief Title: A Study in Adult Patients With Type I, III or IV Osteogenesis Imperfecta Treated With BPS804
Acronym: Asteroid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBPS205; 2016-005096-27 (EudraCT Number)
Record Dates: First submitted 2017-04-03; First posted 2017-04-18 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2022-02

CONDITIONS: Osteogenesis Imperfecta, Type I; Osteogenesis Imperfecta Type III; Osteogenesis Imperfecta Type IV
Keywords: Osteogenesis Imperfecta; Brittle Bone Disease
MeSH Terms: conditions — Osteogenesis Imperfecta; Osteogenesis imperfecta, type 3 | interventions — setrusumab; Calcium; Vitamin D; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: Double-blind, Dose-finding Study, incorporating an open-label substudy
Who Masked: Participant, Investigator
Masking Description: Sponsor will be masked until the primary analysis of the study except for open-label substudy treatment arm. The study site pharmacist will be unmasked to treatment allocation throughout. Study treatment will be monitored by a separate unmasked monitoring team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Setrusumab 20 mg/kg (Blinded) (Experimental): Setrusumab 20 mg/kg intravenous (IV) infusion once a month for 12 months plus 500 mg calcium oral tablets and 800 IU vitamin D capsules.
  Interventions: Drug: setrusumab; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D; Drug: zoledronic acid (optional)
- Setrusumab 8 mg/kg (Blinded) (Experimental): Setrusumab 8 mg/kg IV infusion once a month for 12 months plus 500 mg calcium oral tablets and 800 IU vitamin D capsules.
  Interventions: Drug: setrusumab; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D; Drug: zoledronic acid (optional)
- Setrusumab 2 mg/kg (Blinded) (Experimental): Setrusumab 2 mg/kg IV infusion once a month for 12 months plus 500 mg calcium oral tablets and 800 IU vitamin D capsules.
  Interventions: Drug: setrusumab; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D; Drug: zoledronic acid (optional)
- Setrusumab 20 mg/kg (Open-Label) (Experimental): Setrusumab 20 mg/kg IV infusion once a month for 12 months plus 500 mg calcium oral tablets and 800 IU vitamin D capsules.
  Interventions: Drug: setrusumab; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D; Drug: zoledronic acid (optional)
- Placebo (Placebo Comparator): Placebo IV infusion once a month for 12 months plus 500 mg calcium oral tablets and 800 IU vitamin D capsules.
  Interventions: Dietary Supplement: Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: setrusumab — Intravenous infusion
  Other Names: BPS804
  Arms: Setrusumab 2 mg/kg (Blinded); Setrusumab 20 mg/kg (Blinded); Setrusumab 20 mg/kg (Open-Label); Setrusumab 8 mg/kg (Blinded)
Dietary Supplement: Calcium — tablets
Dietary Supplement: Vitamin D — capsules
Drug: zoledronic acid (optional) — Following completion of the study treatment (Month 12) participants can receive an optional single dose of zoledronic acid. Participants can receive an optional further dose of zoledronic acid at Month 18 at the discretion of their treating physician.
  Arms: Setrusumab 2 mg/kg (Blinded); Setrusumab 20 mg/kg (Blinded); Setrusumab 20 mg/kg (Open-Label); Setrusumab 8 mg/kg (Blinded)

SUMMARY:
The purpose of this study is to select a suitable dose of BPS804 by measuring the strength/quality of bone using a special type of CT scanner. Participants will be treated for 12 months and followed up for a further 12 months.

DETAILED DESCRIPTION:
This study was previously posted by Mereo Biopharma and was transferred to Ultragenyx in February 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of OI Type I, III or IV with a confirmed defect in the COL1A1/COL1A2 genes, as confirmed by genetic testing
* One or more fractures in the past 5 years
* Capable of giving signed consent

Exclusion Criteria:

* History of skeletal malignancies or other bone diseases (other than OI)
* History of neural foraminal stenosis (except if due to scoliosis)
* History of myocardial infarction, angina pectoris, ischaemic stroke or transient ischaemic attack
* History of endocrine or thyroid/parathyroid conditions that could affect bone metabolism
* Treatment with bisphosphonates within 3 months of randomisation
* Treatment with teraparatide, denosumab or other anabolic/anti-reabsorptive medications within 6 months of randomisation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Mereo BioPharma
Locations (25):
- United States (12):
  - Mereo Investigator Site, Birmingham, Alabama
  - Mereo Investigator Site, Jacksonville, Florida
  - Mereo Investigator Site, Baltimore, Maryland
  - Mereo Investigator Site, Boston, Massachusetts
  - Mereo Investigator Site, Saint Paul, Minnesota
  - Mereo Investigator Site, St Louis, Missouri
  - Mereo Investigator Site, Albuquerque, New Mexico
  - Mereo Investigator Site, Cincinnati, Ohio
  - Mereo Investigator Site, Portland, Oregon
  - Mereo Investigator Site, Pittsburgh, Pennsylvania
  - Mereo Investigator Site, Nashville, Tennessee
  - Mereo Investigator Site, Houston, Texas
- Canada (3):
  - Mereo Investigator Site, Toronto, Ontario
  - Mereo Investigator Site, Montreal, Quebec
  - Mereo Investigator Site, Québec, Quebec
- Denmark (2):
  - Mereo Investigator Site, Aarhus
  - Mereo Investigator Site, Odense
- France (3):
  - Mereo Investigator Site, Paris, Paris Cedex 14
  - Mereo Investigator Site, Lyon
  - Mereo Investigator Site, Paris
- United Kingdom (5):
  - Mereo Investigator Site, Cambridge, Cambridgeshire
  - Mereo Investigator Site, Newcastle upon Tyne, Newcastle
  - Mereo Investigator Site, Oxford, Oxfordshire
  - Mereo Investigator Site, Bristol
  - Mereo Investigator Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized 1:1:1:1 to 3 doses of setrusumab (20 mg/kg, 8 mg/kg and 2 mg/kg) and placebo for a 12-month Treatment Period. Per Protocol Amendment 4, participants originally randomized to the placebo group were reassigned to receive 20 mg/kg open-label setrusumab (1 discontinued study prior to the transition). Two participants in the setrusumab 20 mg/kg open-label group were randomized into this group after Amendment 4 and did not receive placebo.
Groups:
- Setrusumab 20 mg/kg (Open-Label): Setrusumab 20 mg/kg IV infusion once a month for 12 months plus 500 mg calcium oral tablets and 800 IU vitamin D capsules. Participants were randomized to this group after amendment 4.
- Placebo: Placebo IV infusion once a month for 12 months plus 500 mg calcium oral tablets and 800 IU vitamin D capsules. Due to a protocol amendment, placebo was actually received for an average of 5 months. Participants originally randomized to the placebo group were reassigned to receive 20 mg/kg open-label setrusumab after amendment 4.
Period: Overall Study
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded) | Setrusumab 20 mg/kg (Open-Label) | Placebo
Started | 31 | 29 | 30 | 2 | 20
Reassigned From Placebo to 20 mg/kg Open-Label Setrusumab | 0 | 0 | 0 | 0 | 19
Completed | 26 | 22 | 25 | 2 | 15
Not Completed | 5 | 7 | 5 | 0 | 5
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 4 | 0 | 1
Not completed — Lost to Follow-up | 2 | 3 | 1 | 0 | 1
Not completed — Other, Not Specified | 1 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 19 participants who transitioned from the Placebo arm to the Setrusumab 20 mg/kg Open-Label arm are NOT "double-counted" for this analysis.
Groups:
- Setrusumab 20 mg/kg (Blinded); Setrusumab 20 mg/kg (Open-Label): Setrusumab 20 mg/kg IV infusion once a month for 12 months plus 500 mg calcium oral tablets and 800 IU vitamin D capsules.
- Placebo: Placebo IV infusion once a month for 12 months plus 500 mg calcium oral tablets and 800 IU vitamin D capsules. Due to a protocol amendment, placebo was actually received for an average of 5 months.
- Total: Total of all reporting groups
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded) | Setrusumab 20 mg/kg (Open-Label) | Placebo | Total
Number analyzed (Participants) | 31 | 29 | 30 | 2 | 20 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (13.73) | 40.4 (14.34) | 47.2 (12.42) | 43.5 (14.85) | 40.9 (14.68) | 42.4 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 21 | 1 | 14 | 73
  Male | 14 | 9 | 9 | 1 | 6 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 0 | 1 | 7
  Not Hispanic or Latino | 27 | 27 | 28 | 2 | 19 | 103
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 1 | 1 | 0 | 0 | 4
  White | 29 | 27 | 29 | 2 | 20 | 107
  Not Collected or Not Reported | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Radial Trabecular Volumetric Bone Mineral Density (Tr vBMD) at Month 12
Description: Assessed by high resolution peripheral quantitative computed tomography (HRpQCT). HRpQCT scans were performed on the participant's distal non-dominant arm. In cases of an arm that had been supported with rods or had significant deformity, the dominant limb was selected. Data presents the ratio of the means between the visit and Baseline from analysis of covariance (ANCOVA).
Time Frame: Baseline, Month 12 (end of treatment [EOT])
Population: Full Analysis Set: all participants who are randomized to one of the blinded treatment arms and took at least 1 dose of study treatment (per protocol almost all efficacy endpoints were to be analyzed only in the blinded treatment arms). Participants with an assessment at given time point.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
ratio | 1.004 [0.987 to 1.021] | 0.993 [0.975 to 1.012] | 0.992 [0.974 to 1.011]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.644, ANCOVA — Analysis is based on a log transformed analysis of covariance (ANCOVA) model with change from baseline as outcome parameter; including categorical effects of treatment and randomization stratum as well as the associated baseline value as a covariate
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.485, ANCOVA — Analysis is based on a log transformed ANCOVA model with change from baseline as outcome parameter; including categorical effects of treatment and randomization stratum as well as the associated baseline value as a covariate
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.404, ANCOVA — [p-value comment as in outcome 1, analysis 2]

2. Primary Outcome: Change From Baseline in Radial Bone Strength (Failure Load) at Month 12
Description: Assessed by finite element analysis (FEA) of models generated from HRpQCT images of the distal radius.
Time Frame: Baseline, Month 12 (EOT)
Population: Full Analysis Set: all participants who are randomized to one of the blinded treatment arms and took at least 1 dose of study treatment. Participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: newton (N)
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 28 | 22 | 25
newton (N) | 61.25 (21.669) | 32.25 (24.342) | 8.86 (23.200)
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.006, ANCOVA — Analysis is based on an ANCOVA model with Change from Baseline as outcome parameter; including categorical effects of treatment and randomization stratum as well as the associated baseline value as a covariate
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.190, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.704, ANCOVA — [p-value comment as in outcome 2, analysis 1]

3. Primary Outcome: Change From Baseline in Radial Bone Strength (Stiffness) at Month 12
Description: Assessed by FEA of models generated from HRpQCT images of the distal radius.
Time Frame: Baseline, Month 12 (EOT)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: N/mm
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 28 | 22 | 25
N/mm | 1638.70 (625.808) | 1422.00 (703.275) | 209.89 (671.777)
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.011, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.047, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.756, ANCOVA — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Radial and Tibial Tr VBMD Over Time: Full Analysis Set
Description: Assessed by HRpQCT. HRpQCT scans were performed on the participant's distal non-dominant arm. In cases of an arm that had been supported with rods or had significant deformity, the dominant limb was selected. Data presented is the ratio of the means between the Visit and Baseline from ANCOVA.
Time Frame: Baseline, Months 6, 12 (EOT), 18, 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
ratio
  Radial: Month 6: number analyzed (Participants) | 26 | 25 | 25
  Radial: Month 6 | 1.007 [0.993 to 1.021] | 1.000 [0.986 to 1.015] | 0.998 [0.984 to 1.013]
  Radial: Month 12: number analyzed (Participants) | 28 | 22 | 24
  Radial: Month 12 | 1.004 [0.987 to 1.021] | 0.993 [0.975 to 1.012] | 0.992 [0.974 to 1.011]
  Radial: Month 18: number analyzed (Participants) | 23 | 17 | 23
  Radial: Month 18 | 1.002 [0.984 to 1.020] | 0.992 [0.973 to 1.013] | 0.979 [0.962 to 0.997]
  Radial: Month 24: number analyzed (Participants) | 21 | 16 | 16
  Radial: Month 24 | 0.997 [0.972 to 1.023] | 0.998 [0.970 to 1.027] | 0.979 [0.951 to 1.008]
  Tibial: Month 6: number analyzed (Participants) | 23 | 20 | 17
  Tibial: Month 6 | 1.004 [0.986 to 1.022] | 1.016 [0.996 to 1.036] | 0.990 [0.969 to 1.012]
  Tibial: Month 12: number analyzed (Participants) | 24 | 17 | 15
  Tibial: Month 12 | 0.991 [0.940 to 1.046] | 1.018 [0.955 to 1.086] | 0.973 [0.909 to 1.042]
  Tibial: Month 18: number analyzed (Participants) | 20 | 13 | 16
  Tibial: Month 18 | 0.989 [0.945 to 1.035] | 1.042 [0.985 to 1.102] | 0.983 [0.933 to 1.036]
  Tibial: Month 24: number analyzed (Participants) | 19 | 12 | 11
  Tibial: Month 24 | 1.000 [0.949 to 1.054] | 1.062 [0.995 to 1.133] | 1.017 [0.949 to 1.090]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.329, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.953, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.795, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.644, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.485, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.404, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.827, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.459, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.022, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.821, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.911, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.152, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.668, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.109, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.358, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.742, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.567, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.430, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.634, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.146, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.521, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.991, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.069, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.625, ANCOVA — [p-value comment as in outcome 1, analysis 2]

5. Secondary Outcome: Changes From Baseline in Radial and Tibial Tr VBMD at Months 6 and 12: Open-Label Arm
Description: as for outcome 4
Time Frame: Baseline, Months 6, 12 (EOT)
Population: All participants in the open-label arm who took at least 1 dose of study treatment. Participants with an assessment at given time point.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Setrusumab 20 mg/kg (Open-Label)
Number analyzed (Participants) | 21
ratio
  Radial: Month 6: number analyzed (Participants) | 17
  Radial: Month 6 | 0.994 [0.972 to 1.017]
  Radial: Month 12: number analyzed (Participants) | 16
  Radial: Month 12 | 1.011 [0.986 to 1.036]
  Tibial: Month 6: number analyzed (Participants) | 15
  Tibial: Month 6 | 1.013 [0.991 to 1.035]
  Tibial: Month 12: number analyzed (Participants) | 15
  Tibial: Month 12 | 1.035 [0.975 to 1.099]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Open-Label); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.615, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Setrusumab 20 mg/kg (Open-Label); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.376, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Setrusumab 20 mg/kg (Open-Label); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.259, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Open-Label); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.253, ANCOVA — [p-value comment as in outcome 1, analysis 2]

6. Secondary Outcome: Changes From Baseline in Radial and Tibial Bone Strength (Failure Load) Over Time: Full Analysis Set
Description: Assessed by FEA of models generated from HRpQCT images of the distal radius.
Time Frame: Baseline, Months 6, 12 (EOT), 18, 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: N
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
N
  Radial: Month 6: number analyzed (Participants) | 26 | 25 | 26
  Radial: Month 6 | 31.22 [-1.80 to 64.23] | 39.95 [6.63 to 73.27] | -3.28 [-36.57 to 30.00]
  Radial: Month 12: number analyzed (Participants) | 28 | 22 | 25
  Radial: Month 12 | 61.25 [18.03 to 104.46] | 32.25 [-16.30 to 80.80] | 8.86 [-37.41 to 55.13]
  Radial: Month 18: number analyzed (Participants) | 23 | 17 | 24
  Radial: Month 18 | 50.39 [19.11 to 81.68] | 43.11 [6.79 to 79.42] | -10.53 [-41.86 to 20.80]
  Radial: Month 24: number analyzed (Participants) | 21 | 16 | 17
  Radial: Month 24 | -19.59 [-72.66 to 33.47] | 45.03 [-14.40 to 104.47] | -50.65 [-108.69 to 7.39]
  Tibial: Month 6: number analyzed (Participants) | 23 | 20 | 17
  Tibial: Month 6 | 46.00 [-24.91 to 116.92] | 45.91 [-28.16 to 119.98] | -65.33 [-146.39 to 15.72]
  Tibial: Month 12: number analyzed (Participants) | 24 | 17 | 15
  Tibial: Month 12 | 76.15 [-11.23 to 163.54] | 60.20 [-42.63 to 163.04] | -65.96 [-175.43 to 43.51]
  Tibial: Month 18: number analyzed (Participants) | 20 | 13 | 16
  Tibial: Month 18 | 50.69 [-34.55 to 135.93] | 88.33 [-13.67 to 190.32] | -49.50 [-144.93 to 45.94]
  Tibial: Month 24: number analyzed (Participants) | 19 | 12 | 11
  Tibial: Month 24 | -24.75 [-126.76 to 77.27] | 41.37 [-86.68 to 169.43] | -74.94 [-208.22 to 58.34]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.064, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.019, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.845, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.006, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.190, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.704, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.002, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.021, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.504, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.462, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.134, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.086, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.199, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 8; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.219, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.112, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.086, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.245, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.232, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.237, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.088, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.302, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.626, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 8; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.517, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.262, ANCOVA — [p-value comment as in outcome 2, analysis 1]

7. Secondary Outcome: Changes From Baseline in Radial and Tibial Bone Strength (Failure Load) at Months 6 and 12: Open-Label Arm
Description: Assessed by FEA of models generated from HRpQCT images of the distal radius.
Time Frame: Baseline, Months 6, 12 (EOT)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: N
Arm/Group | Setrusumab 20 mg/kg (Open-Label)
Number analyzed (Participants) | 21
N
  Radial: Month 6: number analyzed (Participants) | 16
  Radial: Month 6 | 110.16 [61.30 to 159.01]
  Radial: Month 12: number analyzed (Participants) | 15
  Radial: Month 12 | 88.32 [28.55 to 148.09]
  Tibial: Month 6: number analyzed (Participants) | 15
  Tibial: Month 6 | 69.78 [-8.61 to 148.18]
  Tibial: Month 12: number analyzed (Participants) | 15
  Tibial: Month 12 | 112.92 [10.76 to 215.07]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Open-Label); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 20 mg/kg (Open-Label); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.004, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 20 mg/kg (Open-Label); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.080, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Open-Label); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.031, ANCOVA — [p-value comment as in outcome 2, analysis 1]

8. Secondary Outcome: Changes From Baseline in Radial and Tibial Bone Strength (Stiffness) Over Time: Full Analysis Set
Description: Assessed by FEA of models generated from HRpQCT images of the distal radius.
Time Frame: Baseline, Months 6, 12 (EOT), 18, 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: N/mm
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
N/mm
  Radial: Month 6: number analyzed (Participants) | 26 | 25 | 26
  Radial: Month 6 | 795.67 [-34.71 to 1626.04] | 1048.61 [209.47 to 1887.75] | 109.65 [-728.52 to 947.82]
  Radial: Month 12: number analyzed (Participants) | 28 | 22 | 25
  Radial: Month 12 | 1638.70 [390.57 to 2886.83] | 1422.00 [19.37 to 2824.64] | 209.89 [-1129.93 to 1549.71]
  Radial: Month 18: number analyzed (Participants) | 23 | 17 | 24
  Radial: Month 18 | 1295.98 [390.54 to 2201.42] | 803.50 [-263.21 to 1870.21] | -215.92 [-1132.78 to 700.94]
  Radial: Month 24: number analyzed (Participants) | 21 | 16 | 17
  Radial: Month 24 | -625.46 [-1888.53 to 637.60] | 1172.45 [-265.87 to 2610.76] | -1258.55 [-2663.69 to 146.60]
  Tibial: Month 6: number analyzed (Participants) | 23 | 20 | 17
  Tibial: Month 6 | 1344.84 [-296.83 to 2986.52] | 1051.40 [-708.46 to 2811.25] | -1356.71 [-3284.14 to 570.73]
  Tibial: Month 12: number analyzed (Participants) | 24 | 17 | 15
  Tibial: Month 12 | 2326.63 [221.71 to 4431.55] | 1543.85 [-973.70 to 4061.40] | -1428.87 [-4118.78 to 1261.03]
  Tibial: Month 18: number analyzed (Participants) | 20 | 13 | 16
  Tibial: Month 18 | 1047.16 [-1070.79 to 3165.11] | 1697.21 [-861.80 to 4256.23] | -815.38 [-3247.85 to 1617.09]
  Tibial: Month 24: number analyzed (Participants) | 19 | 12 | 11
  Tibial: Month 24 | -1250.69 [-4131.64 to 1630.26] | 622.77 [-2966.46 to 4212.01] | -1844.84 [-5695.04 to 2005.37]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.060, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.015, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.795, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.011, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.047, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.756, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.006, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.137, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.639, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.325, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.108, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.078, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.106, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.236, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.164, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.031, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.224, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.291, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.324, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.188, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.503, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.385, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.727, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.338, ANCOVA — [p-value comment as in outcome 2, analysis 1]

9. Secondary Outcome: Changes From Baseline in Radial and Tibial Bone Strength (Stiffness) at Months 6 and 12: Open-Label Arm
Description: Assessed by FEA of models generated from HRpQCT images of the distal radius.
Time Frame: Baseline, Months 6, 12 (EOT)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: N/mm
Arm/Group | Setrusumab 20 mg/kg (Open-Label)
Number analyzed (Participants) | 21
N/mm
  Radial: Month 6: number analyzed (Participants) | 16
  Radial: Month 6 | 5056.51 [3404.58 to 6708.45]
  Radial: Month 12: number analyzed (Participants) | 15
  Radial: Month 12 | 4992.82 [3056.80 to 6928.84]
  Tibial: Month 6: number analyzed (Participants) | 15
  Tibial: Month 6 | 4225.92 [1840.16 to 6611.68]
  Tibial: Month 12: number analyzed (Participants) | 15
  Tibial: Month 12 | 5827.81 [2601.54 to 9054.08]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Open-Label); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 20 mg/kg (Open-Label); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 20 mg/kg (Open-Label); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Open-Label); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

10. Secondary Outcome: Percentage of Participants With at Least 1 New Fracture (Peripheral, Vertebral, Long-Bone, Any) at Month 12
Description: Fracture assessment, confirmed by central radiographic reading, was carried out for peripheral including all major long bones, minor bone (digits, ribs) and vertebral fractures. Fractures without clinical symptoms, detected only by means of radiographic investigations, were not included in the analysis.
Time Frame: Month 12 (EOT)
Population: Full Analysis Set: all participants who are randomized to one of the blinded treatment arms and took at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
percentage of participants
  Peripheral | 6.5 | 17.2 | 13.3
  Vertebral | 0 | 0 | 0
  Long-Bone | 3.2 | 13.8 | 3.3
  Any | 16.1 | 34.5 | 23.3

11. Secondary Outcome: Change From Baseline in Lumbar, Total Body, and Femoral Neck Bone Mineral Density (BMD) T-score at Month 6
Description: BMD was evaluated by dual-energy x-ray absorptiometry (DXA). T-Score was calculated based on actual measured bone density value. T-scores are standardized scores that reflect the standard deviations (SDs) above/below the normal mean for young adults. A score of 50 indicates the population mean with a standard deviation of 10. A positive change in DXA T-score indicates an improvement in BMD.
Time Frame: Baseline, Month 6
Population: Full Analysis Set: all participants who are randomized to one of the blinded treatment arms and took at least 1 dose of study treatment. Participants with an assessment at given timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
T-score
  Lumbar: number analyzed (Participants) | 24 | 25 | 26
  Lumbar | 0.273 [0.142 to 0.405] | 0.338 [0.213 to 0.464] | 0.110 [-0.014 to 0.233]
  Total Body: number analyzed (Participants) | 23 | 24 | 27
  Total Body | 0.072 [-0.049 to 0.194] | 0.071 [-0.048 to 0.189] | 0.122 [0.009 to 0.235]
  Femoral Neck: number analyzed (Participants) | 21 | 19 | 24
  Femoral Neck | -0.024 [-0.143 to 0.095] | 0.102 [-0.023 to 0.226] | 0.087 [-0.026 to 0.199]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.080, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.238, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.238, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.035, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.687, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.107, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.128, ANCOVA — [p-value comment as in outcome 2, analysis 1]

12. Secondary Outcome: Change From Baseline in Lumbar, Total Body, and Femoral Neck BMD at Month 6
Description: BMD was evaluated by DXA.
Time Frame: Baseline, Month 6
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
g/cm^2
  Lumbar: number analyzed (Participants) | 24 | 25 | 26
  Lumbar | 4.06 [2.12 to 6.00] | 4.70 [2.86 to 6.55] | 1.58 [-0.24 to 3.40]
  Total Body: number analyzed (Participants) | 23 | 24 | 27
  Total Body | 0.77 [-0.38 to 1.92] | 0.83 [-0.29 to 1.94] | 1.21 [0.14 to 2.28]
  Femoral Neck: number analyzed (Participants) | 21 | 19 | 24
  Femoral Neck | -0.42 [-2.51 to 1.68] | 1.64 [-0.57 to 3.84] | 1.61 [-0.38 to 3.59]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.088, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.184, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.144, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.028, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.694, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.143, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.111, ANCOVA — [p-value comment as in outcome 2, analysis 1]

13. Secondary Outcome: Change From Baseline in Lumbar, Total Body, and Femoral Neck BMD T-score at Month 12
Description: BMD was evaluated by DXA. T-Score was calculated based on actual measured bone density value. T-scores are standardized scores that reflect the standard deviations (SDs) above/below the normal mean for young adults. A score of 50 indicates the population mean with a standard deviation of 10. A positive change in DXA T-score indicates an improvement in BMD.
Time Frame: Baseline, Month 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
T-score
  Lumbar: number analyzed (Participants) | 24 | 22 | 25
  Lumbar | 0.587 [0.427 to 0.746] | 0.486 [0.324 to 0.648] | 0.174 [0.022 to 0.327]
  Total Body: number analyzed (Participants) | 23 | 22 | 26
  Total Body | 0.181 [0.051 to 0.310] | 0.199 [0.068 to 0.330] | 0.108 [-0.015 to 0.231]
  Femoral Neck: number analyzed (Participants) | 21 | 18 | 22
  Femoral Neck | 0.163 [0.008 to 0.319] | 0.159 [-0.007 to 0.326] | 0.104 [-0.053 to 0.260]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.026, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.007, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.004, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.085, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.040, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.061, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.189, ANCOVA — [p-value comment as in outcome 2, analysis 1]

14. Secondary Outcome: Change From Baseline in Lumbar, Total Body, and Femoral Neck BMD at Month 12
Description: BMD was evaluated by DXA.
Time Frame: Baseline, Month 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
g/cm^2
  Lumbar: number analyzed (Participants) | 24 | 22 | 25
  Lumbar | 8.55 [6.13 to 10.97] | 6.79 [4.34 to 9.25] | 2.50 [0.19 to 4.81]
  Total Body: number analyzed (Participants) | 23 | 22 | 26
  Total Body | 1.98 [0.70 to 3.25] | 2.03 [0.73 to 3.33] | 1.06 [-0.16 to 2.27]
  Femoral Neck: number analyzed (Participants) | 21 | 18 | 22
  Femoral Neck | 3.30 [0.64 to 5.96] | 2.65 [-0.20 to 5.51] | 1.90 [-0.77 to 4.56]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Lumbar; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.035, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.003, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.003, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Total body; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.088, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.016, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.068, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Femoral neck; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.160, ANCOVA — [p-value comment as in outcome 2, analysis 1]

15. Secondary Outcome: Change From Baseline in Total vBMD (Radial and Tibial) Over Time
Description: as for outcome 4
Time Frame: Baseline, Months 6, 12 (EOT), 18, and 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
ratio
  Radial, Month 6: number analyzed (Participants) | 26 | 25 | 26
  Radial, Month 6 | 1.011 [0.999 to 1.022] | 0.995 [0.984 to 1.007] | 1.000 [0.989 to 1.012]
  Radial, Month 12: number analyzed (Participants) | 28 | 22 | 25
  Radial, Month 12 | 1.017 [1.006 to 1.029] | 1.008 [0.995 to 1.021] | 0.999 [0.986 to 1.011]
  Radial, Month 18: number analyzed (Participants) | 23 | 17 | 24
  Radial, Month 18 | 1.013 [1.000 to 1.026] | 0.992 [0.978 to 1.007] | 0.996 [0.983 to 1.009]
  Radial, Month 24: number analyzed (Participants) | 21 | 16 | 17
  Radial, Month 24 | 0.998 [0.984 to 1.012] | 1.009 [0.994 to 1.025] | 0.985 [0.969 to 1.000]
  Tibial, Month 6: number analyzed (Participants) | 23 | 20 | 17
  Tibial, Month 6 | 1.017 [1.001 to 1.033] | 1.011 [0.995 to 1.028] | 0.995 [0.977 to 1.031]
  Tibial, Month 12: number analyzed (Participants) | 24 | 17 | 15
  Tibial, Month 12 | 1.024 [1.004 to 1.045] | 1.011 [0.988 to 1.035] | 0.989 [0.965 to 1.014]
  Tibial, Month 18: number analyzed (Participants) | 20 | 13 | 16
  Tibial, Month 18 | 1.020 [0.997 to 1.045] | 1.021 [0.992 to 1.050] | 0.987 [0.961 to 1.014]
  Tibial, Month 24: number analyzed (Participants) | 19 | 12 | 11
  Tibial, Month 24 | 1.001 [0.982 to 1.021] | 1.025 [1.001 to 1.050] | 0.994 [0.970 to 1.019]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.065, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.405, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.966, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.003, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.229, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.807, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.042, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.283, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.536, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.765, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.247, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.050, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.037, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.174, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.558, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.020, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.346, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.387, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.093, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.156, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.324, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.920, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.040, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.643, ANCOVA — [p-value comment as in outcome 1, analysis 2]

16. Secondary Outcome: Change From Baseline in Cortical vBMD (Radial and Tibial) Over Time
Description: as for outcome 4
Time Frame: Baseline, Months 6, 12 (EOT), 18, and 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
ratio
  Radial, Month 6: number analyzed (Participants) | 26 | 25 | 26
  Radial, Month 6 | 1.004 [0.997 to 1.010] | 1.002 [0.996 to 1.009] | 0.998 [0.992 to 1.005]
  Radial, Month 12: number analyzed (Participants) | 28 | 22 | 25
  Radial, Month 12 | 1.005 [0.998 to 1.012] | 1.003 [0.995 to 1.010] | 1.001 [0.993 to 1.008]
  Radial, Month 18: number analyzed (Participants) | 23 | 17 | 24
  Radial, Month 18 | 1.011 [1.001 to 1.021] | 1.001 [0.989 to 1.012] | 1.007 [0.997 to 1.017]
  Radial, Month 24: number analyzed (Participants) | 21 | 16 | 17
  Radial, Month 24 | 1.011 [0.999 to 1.022] | 1.018 [1.005 to 1.031] | 1.002 [0.989 to 1.015]
  Tibial, Month 6: number analyzed (Participants) | 23 | 20 | 17
  Tibial, Month 6 | 1.012 [1.003 to 1.022] | 0.997 [0.987 to 1.007] | 0.998 [0.987 to 1.008]
  Tibial, Month 12: number analyzed (Participants) | 24 | 17 | 15
  Tibial, Month 12 | 1.017 [1.008 to 1.026] | 1.004 [0.993 to 1.014] | 0.998 [0.987 to 1.009]
  Tibial, Month 18: number analyzed (Participants) | 20 | 13 | 16
  Tibial, Month 18 | 1.024 [1.009 to 1.039] | 1.004 [0.986 to 1.022] | 0.993 [0.976 to 1.009]
  Tibial, Month 24: number analyzed (Participants) | 19 | 12 | 11
  Tibial, Month 24 | 1.020 [1.004 to 1.035] | 1.017 [0.998 to 1.036] | 0.996 [0.976 to 1.017]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.285, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.544, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.615, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.179, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.513, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.849, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.037, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.880, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.153, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Setrusumab 20 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.073, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Setrusumab 8 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.007, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Setrusumab 2 mg/kg (Blinded); Radial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.791, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.010, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.553, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.652, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.482, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.685, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.002, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.672, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 18; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.377, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 22: Comparison: Setrusumab 20 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.015, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Setrusumab 8 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.086, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 24: Comparison: Setrusumab 2 mg/kg (Blinded); Tibial, Month 24; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.712, ANCOVA — [p-value comment as in outcome 1, analysis 2]

17. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Body Height, Weight and Body Mass Index (BMI) at 6 and 12 Months: Full Analysis Set
Time Frame: Baseline, Month 6, Month 12 (EOT)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
Participants
  Month 6: Body Height | 0 | 0 | 0
  Month 6: Weight | 0 | 0 | 0
  Month 6: BMI | 0 | 0 | 0
  Month 12: Body Height | 0 | 0 | 0
  Month 12: Weight | 0 | 0 | 0
  Month 12: BMI | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline in Lean and Fat Body Mass From Whole Body at Months 6 and 12
Description: Lean and fat body mass was evaluated using whole body DXA (including the head).
Time Frame: Baseline, Months 6, 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: grams
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
grams
  Month 6: Lean: number analyzed (Participants) | 23 | 24 | 27
  Month 6: Lean | 519.152 [13.020 to 1025.284] | -410.664 [-903.724 to 82.395] | 168.206 [-306.981 to 643.393]
  Month 12: Lean: number analyzed (Participants) | 23 | 22 | 26
  Month 12: Lean | 867.668 [204.535 to 1530.801] | -225.474 [-901.083 to 450.136] | 184.164 [-448.625 to 816.953]
  Month 6: Fat: number analyzed (Participants) | 23 | 24 | 27
  Month 6: Fat | 42.567 [-771.815 to 856.949] | 105.420 [-676.720 to 887.561] | 426.388 [-326.298 to 1179.074]
  Month 12: Fat: number analyzed (Participants) | 23 | 22 | 26
  Month 12: Fat | 421.266 [-629.870 to 1472.401] | -85.495 [-1136.234 to 965.245] | 792.485 [-191.238 to 1776.208]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Lean, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.045, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Lean, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.101, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Lean, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.482, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Lean, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.011, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Lean, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.508, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Lean, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.563, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Fat, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.917, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Fat, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.789, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Fat, Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.262, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Setrusumab 20 mg/kg (Blinded); Fat, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.426, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Setrusumab 8 mg/kg (Blinded); Fat, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.871, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Setrusumab 2 mg/kg (Blinded); Fat, Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.113, ANCOVA — [p-value comment as in outcome 1, analysis 2]

19. Secondary Outcome: Change From Baseline in Amino-Terminal Propeptide of Type 1 Procollagen (P1NP) up to Month 12
Time Frame: Baseline, Months 1, 3, 6, 9, 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: µg/L
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
µg/L
  Month 1: number analyzed (Participants) | 30 | 27 | 29
  Month 1 | 24.349 [18.604 to 30.095] | 14.288 [8.221 to 20.354] | 0.060 [-5.827 to 5.948]
  Month 3: number analyzed (Participants) | 29 | 27 | 25
  Month 3 | 17.903 [11.412 to 24.395] | 6.735 [0.015 to 13.455] | 0.640 [-6.389 to 7.670]
  Month 6: number analyzed (Participants) | 27 | 28 | 27
  Month 6 | 13.096 [5.468 to 20.725] | 6.665 [-0.788 to 14.118] | -0.429 [-8.116 to 7.258]
  Month 9: number analyzed (Participants) | 27 | 25 | 26
  Month 9 | 7.265 [-0.115 to 14.644] | 0.238 [-7.353 to 7.830] | -2.254 [-9.820 to 5.312]
  Month 12: number analyzed (Participants) | 25 | 20 | 20
  Month 12 | 5.452 [-3.362 to 14.267] | 4.172 [-5.529 to 13.874] | 4.428 [-5.689 to 14.545]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Month 1; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Month 1; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Month 1; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.984, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Month 3; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Month 3; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.050, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Month 3; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.857, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.079, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.912, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Setrusumab 20 mg/kg (Blinded); Month 9; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.054, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Setrusumab 8 mg/kg (Blinded); Month 9; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.950, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: Setrusumab 2 mg/kg (Blinded); Month 9; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.555, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: Setrusumab 20 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.221, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: Setrusumab 8 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.393, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Setrusumab 2 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.385, ANCOVA — [p-value comment as in outcome 2, analysis 1]

20. Secondary Outcome: Change From Baseline in Carboxy-Terminal Telo-Peptide [CTX-1] up to Month 12
Time Frame: Baseline, Months 1, 3, 6, 9, 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: µg/L
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
µg/L
  Month 1: number analyzed (Participants) | 30 | 27 | 29
  Month 1 | -0.077 [-0.100 to -0.054] | -0.047 [-0.071 to -0.022] | -0.041 [-0.064 to -0.017]
  Month 3: number analyzed (Participants) | 29 | 27 | 25
  Month 3 | -0.044 [-0.071 to -0.016] | -0.029 [-0.058 to 0.000] | -0.043 [-0.073 to -0.013]
  Month 6: number analyzed (Participants) | 27 | 28 | 27
  Month 6 | -0.013 [-0.055 to 0.028] | -0.025 [-0.065 to 0.016] | -0.028 [-0.069 to 0.014]
  Month 9: number analyzed (Participants) | 27 | 25 | 26
  Month 9 | -0.020 [-0.067 to 0.026] | -0.039 [-0.087 to 0.009] | -0.031 [-0.079 to 0.017]
  Month 12: number analyzed (Participants) | 25 | 20 | 20
  Month 12 | -0.037 [-0.083 to 0.010] | -0.002 [-0.053 to 0.049] | -0.034 [-0.087 to 0.019]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Month 1; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Month 1; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Month 1; Test type: Superiority — Comparison is between the Visit and Baseline; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Month 3; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.003, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Month 3; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.050, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Month 3; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.006, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Setrusumab 20 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.519, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Setrusumab 8 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.226, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Setrusumab 2 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.190, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Setrusumab 20 mg/kg (Blinded); Month 9; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.388, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Setrusumab 8 mg/kg (Blinded); Month 9; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.109, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: Setrusumab 2 mg/kg (Blinded); Month 9; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.204, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: Setrusumab 20 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.119, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: Setrusumab 8 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.925, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Setrusumab 2 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.204, ANCOVA — [p-value comment as in outcome 2, analysis 1]

21. Secondary Outcome: Change From Baseline in Short Form 12 Health Survey (SF-12) Physical Component Summary Score at Months 6 and 12
Description: The SF-12 is a generic, 12-item survey that measures 8 domains of health: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It yields scale scores for each of these 8 domains and 2 summary measures of physical and mental health: The Physical Component Summary and the Mental Component Summary. The total score for the Physical Component Summary ranges from 0 to 100, where higher scores reflect better physical functioning.
Time Frame: Baseline, Months 6, 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
score on a scale
  Month 6: number analyzed (Participants) | 27 | 29 | 27
  Month 6 | 0.672 [-1.788 to 3.132] | -0.463 [-2.821 to 1.895] | 1.342 [-1.129 to 3.814]
  Month 12: number analyzed (Participants) | 26 | 26 | 26
  Month 12 | -1.178 [-3.698 to 1.341] | -0.994 [-3.488 to 1.501] | 2.171 [-0.352 to 4.695]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.588, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.697, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.283, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.354, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.430, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.091, ANCOVA — [p-value comment as in outcome 2, analysis 1]

22. Secondary Outcome: Change From Baseline in SF-12 Mental Component Summary Score at Months 6 and 12
Description: The SF-12 is a generic, 12-item survey that measures 8 domains of health: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It yields scale scores for each of these 8 domains and 2 summary measures of physical and mental health: The Physical Component Summary and the Mental Component Summary. The total score for the Mental Component Summary ranges from 0 to 100, where higher scores reflect better mental health functioning.
Time Frame: Baseline, Months 6, 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
score on a scale
  Month 6: number analyzed (Participants) | 27 | 29 | 27
  Month 6 | 0.966 [-2.064 to 3.996] | -0.492 [-3.411 to 2.427] | -1.133 [-4.202 to 1.936]
  Month 12: number analyzed (Participants) | 26 | 26 | 26
  Month 12 | 2.807 [-0.216 to 5.831] | -1.473 [-4.457 to 1.511] | -1.664 [-4.694 to 1.366]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.527, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.738, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.465, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.068, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.328, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.277, ANCOVA — [p-value comment as in outcome 2, analysis 1]

23. Secondary Outcome: Change From Baseline in Index (Utility) Score on EuroQol 5-Dimension 5-Level Descriptive System (EQ-5D-5L) Score at Months 6 and 12
Description: The EQ-5D-5L is a standardised measure of health status comprised of a descriptive system of 5 health-related quality of life states (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a Visual Analogue Scale (VAS) of overall health. Each dimension is rated on a 5-point response scale indicating severity of problems, where 1 is "no problems" and 5 is "extreme problems". The 5 questions are scored and together contribute to the EQ-5D index (utility) score between 0 and 1 (1 being perfect health).
Time Frame: Baseline, Months 6 and 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
score on a scale
  Month 6: number analyzed (Participants) | 27 | 28 | 26
  Month 6 | 0.0627 [-0.0105 to 0.1359] | 0.0362 [-0.0343 to 0.1067] | -0.0383 [-0.1121 to 0.0354]
  Month 12: number analyzed (Participants) | 26 | 25 | 26
  Month 12 | 0.0424 [-0.0163 to 0.1012] | 0.0252 [-0.0332 to 0.0837] | 0.0214 [-0.0365 to 0.0793]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.092, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.310, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.304, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.155, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.392, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.464, ANCOVA — [p-value comment as in outcome 2, analysis 1]

24. Secondary Outcome: Change From Baseline in Osteogenesis Imperfecta Specific Quality of Life Questionnaire for Adults (OIQoL-A) Total Score at Months 6 and 12
Description: The OIQoL-A measures 5 areas of quality of life related to OI (Physical Function, Pain, Hearing Loss, Taking Care/Concerns, Social and Family Life and Activities). The total score is calculated on a 0-100 scale, where higher scores indicate a greater (negative) impact on quality of life.
Time Frame: Baseline, Months 6, 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
score on a scale
  Month 6: number analyzed (Participants) | 27 | 25 | 26
  Month 6 | -3.584 [-8.491 to 1.324] | -1.848 [-6.899 to 3.203] | -0.649 [-5.751 to 4.452]
  Month 12: number analyzed (Participants) | 25 | 24 | 25
  Month 12 | -1.668 [-7.395 to 4.059] | -0.587 [-6.310 to 5.137] | -3.846 [-9.592 to 1.901]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.150, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.468, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.800, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.563, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.839, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.186, ANCOVA — [p-value comment as in outcome 2, analysis 1]

25. Secondary Outcome: Change From Baseline in OIQoL-A Pain Subscale Score at Months 6 and 12
Description: The OIQoL-A measures 5 areas of quality of life related to OI (Physical Function, Pain, Hearing Loss, Taking Care/Concerns, Social and Family Life and Activities). The Pain subscale ranges from 0 to 10, with higher value representing worse pain.
Time Frame: Baseline, Months 6, 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
score on a scale
  Month 6: number analyzed (Participants) | 27 | 26 | 26
  Month 6 | -3.990 [-11.267 to 3.287] | -3.906 [-11.239 to 3.426] | -6.003 [-13.495 to 1.489]
  Month 12: number analyzed (Participants) | 26 | 26 | 25
  Month 12 | -3.655 [-11.505 to 4.195] | -4.968 [-12.709 to 2.772] | -7.178 [-15.183 to 0.827]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.278, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.292, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.115, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.356, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.205, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.078, ANCOVA — [p-value comment as in outcome 2, analysis 1]

26. Secondary Outcome: Change From Baseline in OIQoL-A Activity Subscale Score at Months 6 and 12
Description: The OIQoL-A measures 5 areas of quality of life related to OI (Physical Function, Pain, Hearing Loss, Taking Care/Concerns, Social and Family Life and Activities). The Activities subscale ranges from 0 to 100, with higher value representing increased difficulty.
Time Frame: Baseline, Months 6, 12 (EOT)
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded)
Number analyzed (Participants) | 31 | 29 | 30
score on a scale
  Month 6: number analyzed (Participants) | 27 | 26 | 26
  Month 6 | -5.980 [-11.597 to -0.363] | -2.722 [-8.397 to 2.953] | 1.907 [-3.906 to 7.719]
  Month 12: number analyzed (Participants) | 26 | 25 | 25
  Month 12 | -0.964 [-8.006 to 6.079] | 4.489 [-2.620 to 11.598] | -1.630 [-8.869 to 5.609]
Statistical Analysis 1: Comparison: Setrusumab 20 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.037, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Setrusumab 8 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.342, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Setrusumab 2 mg/kg (Blinded); Month 6; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.515, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Setrusumab 20 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.786, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Setrusumab 8 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.212, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Setrusumab 2 mg/kg (Blinded); Month 12; Test type: Superiority — Comparison is between the Visit and Baseline; p = 0.655, ANCOVA — [p-value comment as in outcome 2, analysis 1]

27. Secondary Outcome: Percentage of Participants Who Were Positive for Anti-Setrusumab Antibodies at Any Time During the Study up to Month 14
Description: Serum samples were screened for antibodies binding to setrusumab using a validated assay method by or under the supervision of the sponsor.
Time Frame: up to Month 14
Population: Safety Population: all participants who received at least 1 dose of study drug. The 19 participants who transitioned from the Placebo arm to the Setrusumab 20 mg/kg Open-Label arm are reflected in both arms for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded) | Setrusumab 20 mg/kg (Open-Label) | Placebo
Number analyzed (Participants) | 31 | 29 | 30 | 21 | 20
percentage of participants
  Binding Antibodies | 16.1 | 17.2 | 16.7 | 9.5 | 15.0
  Neutralizing Antibodies | 16.1 | 17.2 | 16.7 | 0 | 0
  Both Binding and Neutralizing Antibodies | 16.1 | 17.2 | 16.7 | 0 | 0

28. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Treatment-Emergent AEs (TEAEs), Serious TEAEs, and TEAEs Leading to Discontinuation or Death
Description: An AE is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment. A serious AE (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; is another important medical event. The intensity for each AE was graded as mild, moderate or severe, according to the investigator's judgement. An event was considered related to study drug if there were a "reasonable possibility" of a relationship, according to the investigator's clinical judgment. A TEAE was defined as an event occurring or worsening on or after the first dose of study medication.
Time Frame: Non-serious AEs: up to Month 14; Serious AEs: up to Month 24. (Average duration of exposure to placebo was 5 months and for setrusumab was 11 month plus follow-up to 24 months.)
Population: as for outcome 27
Measure: Number; unit: percentage of participants
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded) | Setrusumab 20 mg/kg (Open-Label) | Placebo
Number analyzed (Participants) | 31 | 29 | 30 | 21 | 20
percentage of participants
  All AEs | 100.0 | 96.6 | 90.0 | 100.0 | 90.0
  TEAEs | 100.0 | 96.6 | 90.0 | 95.2 | 80.0
  Treatment-Related TEAEs | 71.0 | 41.4 | 36.7 | 42.9 | 25.0
  Serious TEAEs | 12.9 | 24.1 | 23.3 | 23.8 | 10.0
  Treatment-Related Serious TEAEs | 6.5 | 0 | 0 | 9.5 | 0
  TEAEs Leading to Death | 0 | 0 | 0 | 0 | 0
  TEAEs Leading to Permanent Study Treatment Discontinuation | 6.5 | 0 | 0 | 9.5 | 5.0

ADVERSE EVENTS:
Time Frame: Non-serious AEs: up to Month 14; Serious AEs: up to Month 24. (Average duration of exposure to placebo was 5 months and for setrusumab was 11 month plus follow-up to 24 months.)
Description: Safety Population: all participants who received at least 1 dose of study drug. The 19 participants who transitioned from the Placebo arm to the Setrusumab 20 mg/kg Open-Label arm are reflected in both arms for this analysis.
Arm/Group | Setrusumab 20 mg/kg (Blinded) | Setrusumab 8 mg/kg (Blinded) | Setrusumab 2 mg/kg (Blinded) | Setrusumab 20 mg/kg (Open-Label) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 0/30 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 4/31 | 7/29 | 7/30 | 5/21 | 2/20
Other Adverse Events (participants affected / at risk) | 29/31 | 28/29 | 27/30 | 19/21 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Setrusumab 20 mg/kg (Blinded) (N=31) | Setrusumab 8 mg/kg (Blinded) (N=29) | Setrusumab 2 mg/kg (Blinded) (N=30) | Setrusumab 20 mg/kg (Open-Label) (N=21) | Placebo (N=20)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fracture of penis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Joint abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuritis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Platybasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Setrusumab 20 mg/kg (Blinded) (N=31) | Setrusumab 8 mg/kg (Blinded) (N=29) | Setrusumab 2 mg/kg (Blinded) (N=30) | Setrusumab 20 mg/kg (Open-Label) (N=21) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 2 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 2 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 5 | 2 | 2
Toothache (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 3 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 2 | 0
Fatigue (General disorders) | 3 | 2 | 7 | 3 | 0
Influenza like illness (General disorders) | 1 | 2 | 0 | 0 | 0
Injection site extravasation (General disorders) | 1 | 1 | 0 | 1 | 1
Malaise (General disorders) | 0 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 0
Pain (General disorders) | 2 | 0 | 2 | 1 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 2 | 2 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 2 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Ear infection (Infections and infestations) | 3 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 2 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 4 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 3 | 4 | 5 | 3
Sinusitis (Infections and infestations) | 2 | 3 | 4 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 3 | 2 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 4 | 3 | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 3 | 4 | 3 | 6 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 3 | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 3 | 1 | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 3 | 3 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 3 | 2 | 6 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 0 | 0
Aspartate aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 3 | 1 | 1
Lipase increased (Investigations) | 1 | 1 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1 | 3 | 1 | 1
Vitamin D decreased (Investigations) | 0 | 1 | 2 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 8 | 9 | 8 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 8 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 4 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 2 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 3 | 4 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 3 | 0 | 1
Headache (Nervous system disorders) | 4 | 5 | 6 | 7 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT03118570/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT03118570/SAP_001.pdf